CLINICAL TRIAL: NCT02675049
Title: Efficacy and Optimal Dose Selection of Intranasal Dexmedetomidine During Breast Lumpectomy Under Local Anaesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA10
Record Dates: First submitted 2016-01-27; First posted 2016-02-05 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Intranasal Dexmedetomidine Breast Cancer Local Anaesthesia
Keywords: Intranasal; Dexmedetomidine; Anaesthesia; Breast Lumpectomy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.9% saline (Placebo Comparator): Patients were assigned to receive 0.9% saline intranasally 45 min before surgery using a computer-generated random number table.
  Interventions: Drug: 0.9% saline
- dexmedetomidine 1 µg.kg-1 (Experimental): Patients were assigned to receive 1µg.kg-1dexmedetomidine intranasally 45 min before surgery using a computer-generated random number table.
  Interventions: Drug: dexmedetomidine 1µg.kg-1
- dexmedetomidine 1.5 µg.kg-1 (Experimental): Patients were assigned to receive 1.5µg.kg-1 dexmedetomidine intranasally 45 min before surgery using a computer-generated random number table.
  Interventions: Drug: dexmedetomidine 1.5µg.kg-1
- dexmedetomidine 2 µg.kg-1 (Experimental): Patients were assigned to receive 2µg.kg-1 dexmedetomidine intranasally 45 min before surgery using a computer-generated random number table.
  Interventions: Drug: Dexmedetomidine 2µg.kg-1

INTERVENTIONS:
Drug: 0.9% saline — 0.9% saline intranasally 45 min before surgery using a computer-generated random number table.
  Other Names: placebo
  Arms: 0.9% saline
Drug: dexmedetomidine 1µg.kg-1 — dexmedetomidine 1µg.kg-1 intranasally 45 min before surgery using a computer-generated random number table.
  Other Names: Ai Bei Ning1 µg.kg-1
  Arms: dexmedetomidine 1 µg.kg-1
Drug: dexmedetomidine 1.5µg.kg-1 — Dexmedetomidine 1.5µg.kg-1 intranasally 45 min before surgery using a computer-generated random number table.
  Other Names: Ai Bei Ning1 µg.kg-1
  Arms: dexmedetomidine 1.5 µg.kg-1
Drug: Dexmedetomidine 2µg.kg-1 — dexmedetomidine 2µg.kg-1 intranasally 45 min before surgery using a computer-generated random number table.
  Other Names: Ai Bei Ning 2µg.kg-1
  Arms: dexmedetomidine 2 µg.kg-1

SUMMARY:
This trial is going to evaluate the safety and effectiveness of intranasal DEX(dexmedetomidine) in breast lumpectomy under local anaesthesia,and to investigate the optimal dose of intranasal DEX in breast lumpectomy.

DETAILED DESCRIPTION:
Breast lumpectomy associated with a high level of anxiety, fear and pain requires fast and effective anaesthesia techniques. Presently, this procedure is usually performed under general or local anaesthesia. General anaesthesia provides an effective sedation; however, for minor procedures, general anaesthesia is resource-intensive and postoperative complications, such as nausea, vomiting or extended time to ambulation, are more likely. Local anaesthesia alone may be uncomfortable or uncooperative for patients. Therefore, an efficient drug regimen is required that reduces analgesic consumption, minimises opioid-related side effects and shortens post-anaesthesia care unit (PACU) stay following surgery.

Dexmedetomidine (DEX) is a highly selective α2 adrenoreceptor agonist that provides sedation without respiratory depression. Its sedative, anxiolytic, analgesic and haemodynamic effects have made it a useful adjunct to anaesthesia and sedation. DEX may provide a conscious sedation under monitored anaesthesia care (MAC) that is a logical middle ground between general anaesthesia and local anaesthesia. Intranasal DEX was recently shown to provide satisfactory anaesthesia and premedication sedation in healthy volunteers and paediatric patients. The intranasal route is not only effective, but also well-tolerated and convenient This trial is going to evaluate the safety and effectiveness of intranasal DEX(dexmedetomidine) in breast lumpectomy under local anaesthesia, and to investigate the optimal dose of intranasal DEX in breast lumpectomy.

ELIGIBILITY:
Inclusion Criteria:

* with ASA(American Society of Anesthesiologists) physical status I and II
* scheduled for breast lumpectomy

Exclusion Criteria:

* a history of heart block
* upper respiratory tract infection
* asthma
* allergy to DEX or local anaesthetics
* memory or cognitive dysfunction
* pregnancy
* lack of understanding the consent process
* impaired liver or renal function
* a history of drug or alcohol abuse

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Sedation changes using the modified Observer's Assessment of Alertness/Sedation (OAA/S) scale | before surgery,during surgery and after surgery for sedation changes，assessed up to 2 hours
pain scores changes by pain NRS scores | before surgery,during surgery and after surgery for pain scores，assessed up to 2 hours

SECONDARY OUTCOMES:
Adverse event that is related to treatment:severe sinus bradycardia | perioperative period
  bradycardia (defined as HR < 50 bpm)
Adverse event that is related to treatment:hypotension | perioperative period
  hypotension (defined as SBP < 90 mmHg)
Adverse event that is related to treatment:nausea and vomiting | perioperative period

IPD SHARING:
Plan to Share IPD: Undecided